CLINICAL TRIAL: NCT05800288
Title: Clinical Comparison Between Two Propofol TCI Models(Eleveld and Schnider) for General Anaesthesia After Premedication With Midazolam
Brief Title: Effect of Midazolam Bolus on Eleveld and Schnider TCI (Target Controlled Infusion) Models
Acronym: TCI
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Federico Linassi, MD, Principal investigator, University of Padova
Other Study IDs: BenzoMAST
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Propofol; Anesthesia Brain Monitoring
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EleveldTCI: Patients who received Midazolam premedication bolus (0.03 mg/kg) before general anesthesia conducted with Eleveld TCI model (this model was choosen at anesthesiologist's discreption)
  Interventions: Drug: Propofol
- Schnider TCI: Patients who received Midazolam premedication bolus (0.03 mg/kg) before general anesthesia conducted with SchniderTCI model (this model was choosen at anesthesiologist's discreption)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Patients will be observationally included in the Elveld TCI or Schnider TCI group. The TCI model is choosen at anesthesiologist's discreption, as suggested in literature

SUMMARY:
No trials have evaluated the effect of a Midazolam bolus (routinely used for premedication before general anesthesia) on the Concnetration at the effector site of Propofol (CeP) of Eleveld and Schnider TCI models, routinely used for general anesthesia delivery.

DETAILED DESCRIPTION:
During recent years Eleveld and colleagues ideated a new propofol pharmacokinetic/pharmacodynamic (PK/PD) model for total intravenous anaesthesia with target controlled infusion (TIVA-TCI) pumps that has been proposed to have slightly better predictive performance for measured propofol plasma concentrations compared with those of the Marsh and Schnider models, and suitable for children, adults, older subjects, and obese adults, being considered as a "General purpose" model.

However, no trials have compared the Eleveld to the Schnidermodel after a premedication with Midazolam bolus (0.03 mg/kg) from a clinical point of view; so, this study aimed toevaluate midazolam effect on the estimated effector site concentration of the two models (CePE and CePS, respectively) at loss of responsiveness (LoR), during anaesthesia maintenance (Bispectral Index [BIS] 40-60) and return of responsiveness (RoR). The study also compared the incidence of deepening or superficializing anaesthesia (defined respectively as lowering or increasing in out-of-target BIS after initial CeP detection), as well as unwanted anaesthesia events: burst suppression (BSupp, identified as a burst suppression ratio [BSR] >0) and unwanted spontaneous responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Undergo general anaesthsia with Targted Controlld Infusion of Propofol (Eleveld or Schnider model) and Remifentanil (Minto model)after midazolam premedication

Exclusion Criteria:

* Neurological disease
* Psychiatric disease
* Obesity

Ages: 18 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women undergoing brast cancer surgery with general anesthesia with Propofol and Remifentanil TCI, and Midazolam premedication will be recruited
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Concentration at the effector site of Propofol after Midazolam | We will collected data about Drugs concentration and BIS values during general anaesthesia. We will collect BIS and TCI Propofol values during all the duration of anesthesia, form the start of midazolam bolus until the emergence from anesthesia
  Discover if, after astandard premedication with midazolam bolus, there are differences between Concentrations at the effector site of Propofol using the Eleveld TCI model versus Schnider TCI model, during standard general anaesthesia conducted with Propofol and remifenatnil delivered with targeted controlled infusion pumps, usually adopted in our Hospital to delivery general anaesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- ULSS2, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Undecided